CLINICAL TRIAL: NCT02331628
Title: Effect of Extracorporeal Shock Wave Therapy on Chronic Neurogenic Heterotopic Ossification in Traumatic Brain Injured Patients
Brief Title: ESWT as a Treatment for Chronic NHO in TBI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Collaborators: James Cook University, Queensland, Australia (Other); University of Melbourne (Other); Medispec (Industry)
Responsible Party: Principal Investigator, yaron sacher, Yaron Sacher M.D, Loewenstein Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-13
Record Dates: First submitted 2014-12-16; First posted 2015-01-06 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: TBI Traumatic Brain Injury
Keywords: TBI Traumatic Brain Injury; HO Heterotopic Ossification; NHO Neurogenic Heterotopic Ossification; ESWT Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care only will be provided during Baseline period and Follow-up period.
- ESWT - Extracorporeal Shockwave Therapy (Experimental): Participants will receive 4 applications of extracorporeal shockwave therapy to the affected hip and/or knee over a period of 8 weeks (one dose every 2 weeks).
  Interventions: Device: ESWT - Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: ESWT - Extracorporeal Shockwave Therapy — Patients will receive:
  * Four applications of EWST to be delivered to the affected hip and /or knee over a period of eight weeks : starting week 8\52 from baseline until and including week 14\52, one dose every two weeks ± 3 days), administered by the principal investigator.
  * Dosage will be calculated for each participant, by the manufacturer, according to the size of NHO as recorded on X-ray.
  * The energy flux density (EFD) will be 'high level'
  * All participants will be supplied with headphones to reduce the noise level emitted by the machine.
  Other Names: Minispec™ extracorporeal shockwave therapy
  Arms: ESWT - Extracorporeal Shockwave Therapy

SUMMARY:
Effect of Extracorporeal Shock Wave Therapy on Chronic Neurogenic Heterotopic Ossification in Traumatic Brain Injured (TBI) patients

Chronic Neurogenic Heterotopic Ossification (NHO) - Heterotopic ossification is a well known late complication of traumatic brain injury. Extracorporeal Shock Wave Therapy - ESWT- is used in various medical situations and is being tested for feasibility of use in TBI patients.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS Title Effect of Extracorporeal Shock Wave Therapy on Chronic Neurogenic Heterotopic Ossification in Traumatic Brain Injured (TBI) patients.

The investigators primary objective is to determine whether Extracorporeal Shock Wave Therapy (ESWT) is effective in reducing pain and improving function in people with traumatic brain injury who have heterotopic ossification around the hip or knee.

The investigators hypothesize that four applications of ESWT to the affected hip or knee joint in the patient group will demonstrate a positive physiological effect and this will lead to a reduction in pain and improved function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Brain injured patients with a diagnosis of NHO around the hip and/ or knee for a period of greater than one year.
* Patients who are able, or legal guardians who are willing, to provide informed consent after both oral and written information.

Exclusion Criteria:

* Pregnancy.
* Rheumatoid arthritis, ankylosing spondylitis, or femoral neck fractures
* Elevated serum alkaline phosphatase (SAP) levels and/or evidence of active bone remodelling in bone scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (VAS) from baseline to final assessment | VAS will be assessed at two weekly intervals from week 0 (Baseline) until week 22, at week 26 and at week 38.
  The Visual Analogue Pain Scale (VAS) will be used in its format of the Faces Rating Scale (FRS). The FRS is in the format of six facial expressions suggesting various pain intensities. The patient will be asked to choose the face that best describes how they feel. The far left face indicates 'No hurt' and the far right face indicates 'Hurts worst'. The number below the face chosen will be documented.

SECONDARY OUTCOMES:
Change from the 10 Metre Walk at baseline (if patient is ambulatory) | At baseline; weeks 16, 26 and 38
  Temporal and distance measures (velocity, stride length, cadence) will be measured using the 10 metre walk test.
Change from the 6 Minute Walk at baseline (if patient is ambulatory) | At baseline; weeks 16, 26 and 38
  The patient is positioned at the start of the walking track and given the standardized instructions; "Walk as quickly as you can for six minutes to cover as much ground as possible. You may stop if you have to, but continue again as soon as you are able". On the instruction to start the therapist starts the stopwatch. At six minutes the patient is instructed to stop and the distance travelled is calculated. If the patient needs to stop, rest periods are included in the measurement time.
Change from Functional Reach at baseline (if patient is able to stand) | Every two weeks from date of baseline, week 0 up to week 22; then at week 26 and at week 38
  The patient is instructed to stand next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the 3rd metacarpal head on the yardstick. The patient is instructed to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is recorded. The difference between the start and end position is the reach distance, usually measured in centimeters.
  Three trials are done and the average of the last two is noted.
Change from Modified Functional Reach at baseline (if FR not possible) | Every two weeks from date of baseline, week 0 up to week 22; then at week 26 and at week 38
  Modified Functional Reach (MFR) is a reliable measure of sitting balance for those patients unable to stand. This test is performed with a leveled yardstick mounted on the wall at the height of the patient's acromion level while sitting in a chair. Hips, knees and ankles are positioned at 90 degree of flexion, with feet flat on the floor. The initial reach is measured with the patient sitting against the back of the chair with the arm flexed to 90 degrees. The measurement is taken from the distal end of the third metacarpal along the yardstick. There are three conditions over three trials:
  * Sitting with the arm near the wall and leaning forward
  * Sitting with the back to the wall and leaning right
  * Sitting with the back to the wall leaning left. Instructions are leaning as far as possible in each direction without rotation and without touching the wall. The distance in centimetres covered in each direction will be recorded.

OTHER OUTCOMES:
Change from Functional Independence Measure (FIM) at baseline | At baseline; then at 8, 16, 26 and 38 weeks
  The Functional Independence Measure (FIM) assesses physical and cognitive disability. It consists of two subscales, motor and socio-cognitive with 18 assessable items in total. The tool is completed by observation of performance. The motor subscale, which is the portion to be assessed in this trial includes 13 items: eating, grooming bathing, dressing upper extremity, dressing lower extremity, bowel management, bladder management, transfers to bed, chair or wheelchair, transfer to tub, toilet and shower, walking or wheelchair propulsion and stair climbing. Each item is scored on a 7 point ordinal scale ranging from 1 (total dependence) to a score of 7 (total independence). Motor FIM scores range from 13 (total dependence) to 91 (total independence). Reliability and validity is well-established. The FIM has been translated into 10 languages, including English and Hebrew, the languages to be used in this study.
Range of Motion | Every two weeks from week 0 up to week 22; then at weeks 26 and 38
  Range of Motion (ROM) of the affected hip and knee will be measured using a universal goniometer, using the protocol described by Clarkson (2005).
Change from The European Quality Of Life -Dimensions questionnaire (EQ-5D) at baseline | At baseline; 16,26 and 38 weeks
  The European Quality Of Life -Dimensions questionnaire (EQ-5D) is a standardised generic instrument designed for describing and valuing health by providing a single summary index value representing the overall health-related quality of life of an individual by quantifying a preference for his or her health state. The EQ-5D instrument consists of a self-classifier/ descriptive system to describe the respondent's own health in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents can value their health in each dimension at three ordinal levels: no problems, some or moderate problems, and severe or extreme problems. The second measurement component of the EQ-5D is a 20 cm vertical Visual Analogue Scale (EQ VAS) to rate the respondent's own health. The third component of the EQ-5D is a questionnaire on the respondent's background including medical history.
Change from Plain X-ray at baseline | At baseline and six months post first intervention
  Neurogenic Heterotopic Ossification (NHO) becomes evident on plain radiography approximately 2 to 6 weeks after clinical diagnosis (Freed, Hahn, Menter, & Dillon, 1982; Orzel & Rudd, 1985). An X-ray view will be set up for each patient and recorded so that it can be repeated. The view does not need to be a standard view; it is the patient's particular view that is important and reproducible. Measurements will be made along co-ordinates - set up for that patient - e.g. the largest and shortest diameters. Plain X-ray will be taken pre-intervention and six months post-intervention. Changes in the size of NHO will be calculated using UTHSCSA ImageTool (2002).plain radiography .
Change from Serum Alkaline Phosphatase Levels (SAP) at baseline | At base line, week 12, week 16, week 38
  Overview Alkaline Phosphatase Uses Preparation Procedure Risks Results More on Healthline
  Part 1 of 7: Overview What Is an Alkaline Phosphatase Level Test?
  An alkaline phosphatase level test (ALP test) measures the amount of alkaline phosphatase enzyme in your bloodstream. The test requires a simple blood draw and is often a routine part of other blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Sacher, MD, Principal Investigator — Loewenstein Hospital
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel

REFERENCES:
- [Result] Reznik JE, Biros E, Lamont AC, Sacher Y, Kibrik O, Milanese S, Gordon S, Galea MP. A preliminary investigation on the effect of extracorporeal shock wave therapy as a treatment for neurogenic heterotopic ossification following traumatic brain injury. Part I: Effects on pain. Brain Inj. 2017;31(4):526-532. doi: 10.1080/02699052.2017.1283059. Epub 2017 Mar 24. PMID 28340308
- [Result] Reznik JE, Biros E, Sacher Y, Kibrik O, Milanese S, Gordon S, Galea MP. A preliminary investigation on the effect of extracorporeal shock wave therapy as a treatment for neurogenic heterotopic ossification following traumatic brain injury. Part II: Effects on function. Brain Inj. 2017;31(4):533-541. doi: 10.1080/02699052.2017.1283060. Epub 2017 Mar 24. PMID 28340312